CLINICAL TRIAL: NCT05396677
Title: Behavioral Consequences of Blunting Fear With Acetaminophen
Brief Title: The Effects of Acetaminophen on Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Patrick Barclay, Professor of Psychology, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-07-024
Record Dates: First submitted 2022-05-11; First posted 2022-05-31 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Fear
Keywords: acetaminophen; fear; analgesics; virtual reality; emotions
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind placebo study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen Condition (Experimental): 1000 mg acetaminophen
  Interventions: Drug: Acetaminophen
- Placebo Condition (Placebo Comparator): 1000 mg microcrystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetaminophen — 2 x 500 mg acetaminophen (one time)
  Arms: Acetaminophen Condition
Other: Placebo — 2 x 500 mg microcrystalline cellulose (one time)
  Arms: Placebo Condition

SUMMARY:
This study investigates the effects of acetaminophen on behavioral, physiological, and self-report fear responses.

DETAILED DESCRIPTION:
As acetaminophen blunts the experience of physical, social, and empathic pain, it is important to investigate whether there are other aversive states that the drug also provides relief from. If there are others, this may suggest overlapping mechanisms involved in these affective evaluations, all of which are interrupted by acetaminophen. The emotion of fear is aversive, yet it is distinct from both physical and social pain.

The present study will investigate the effects of acetaminophen on the subjective experience of fear as well as its behavioral outcomes. While blocking adaptive behavioral responses to fear could potentially be problematic in some dangerous situations, it may also be helpful for those with anxiety-related disorders. If individuals on acetaminophen can step farther away from safety on a virtual plank 80 stories above the ground, then perhaps acetaminophen can allow anxious individuals to step farther from their comfort zone in real life. Importantly, if acetaminophen blunts the fear response, this would mean that the drug blocks aversive feelings beyond emotional and physical pain. The extent of its effects will warrant further investigation for a greater understanding of emotional evaluations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Literate
* Speaks English
* Does not have any risk factors associated with acetaminophen (history of liver or kidney disease, taking other products with acetaminophen, has any allergies to acetaminophen, taking blood-thinning medications, drinks more than 12 alcoholic drinks per week for females, or more than 15 alcoholic drinks per week for males, are/ could be pregnant)
* Has taken acetaminophen in the past without any adverse reactions
* Is not diabetic
* Did not have anything to eat within three hours of study time
* Did not have any acetaminophen or alcohol in the 48 hours prior to study
* Has never had an adverse reaction to virtual reality before, such as headaches or nausea

Exclusion Criteria:

* Younger than 18
* Non-literate
* Does not speak English
* Has at least one risk factor associated with acetaminophen (history of liver or kidney disease, taking other products with acetaminophen, has any allergies to acetaminophen, taking blood-thinning medications, drinks more than 12 alcoholic drinks per week for females, or more than 15 alcoholic drinks per week for males, are/ could be pregnant)
* Has never taken acetaminophen before
* Diabetic
* Had something to eat within three hours of scheduled study time
* Has had acetaminophen or alcohol in the past 48 hours
* Has had an adverse reaction to virtual reality in the past, such as headaches or nausea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Walking speed on plank in virtual reality | 1 hour after taking acetaminophen or placebo
  Farthest distance reached on plank / time to get there
Distance walked on plank | 1 hour after taking acetaminophen or placebo
  (Unless there are ceiling effects in which >90% of people make it to the end.) Measured in cm walked on a 2 m wooden plank before deciding to turn around and walk back.
Proportion of time spent looking down at the plank | 1 hour after taking acetaminophen or placebo
  We will record what participants see in virtual reality while doing the plank walk, and then code the footage to calculate the proportion of time on the plank participants spent looking down at the plank (indicating more anxiety about falling off).
Decision on whether to do the plank walk again with virtual spiders | 1 hour after taking acetaminophen or placebo
  After doing the plank walk, participants will be offered an optional second chance to try the same plank walk again but this time with virtual giant spiders around them.
Verbal Self-Report Fear | 1 hour after taking acetaminophen or placebo
  While participants are in virtual reality, we will ask them to rate their fear verbally twice, once when they first step onto the plank, and once when they have changed direction (during which the plank tends to shake). They will answer from 0 (no fear or anxiety) to 10 (extreme fear or anxiety). For those who decide to do the plank walk again with virtual giant spiders, they will also rate their self-reported fear in the same manner twice, once when the spiders first appear, and once when they are on their way back to the virtual elevator while surrounded by giant spiders.
Written Self-Report Fear | 1 hour after taking acetaminophen or placebo
  After taking off the headset, participants will answer two survey questions. The first is, "How scary do you think most people would agree the act of walking on a virtual plank is?" They will answer on an 11-point scale (0 = Not at all scary, 5 = Moderately scary, 10 = Extremely scary). They will also be asked "How fearful, scared, nervous, or anxious did you personally feel when walking on the virtual plank?" (0 = Not at all fearful or anxious, 5 = Moderately fearful or anxious, 10 = Extremely fearful or anxious). Those who choose to do the second optional plank walk with virtual spiders will answer the same questions about that experience afterwards.
Heart rate | 1 hour after taking acetaminophen or placebo
  Average heart rate while on the plank walk, measured with a Polar Verity Sense optical heart rate sensor on forearm.

SECONDARY OUTCOMES:
Time to take first step onto plank | 1 hour after taking acetaminophen or placebo
  Number of seconds it takes participants to leave the virtual elevator for the plank overlooking a virtual 80-story drop.
Speed towards virtual elevator after turning around on plank, | 1 hour after taking acetaminophen or placebo
  Amount of time it takes them to make it back to the starting point after turning around on the plank. It is not clear whether someone who walks faster would be doing so to get back to the feeling safety quicker or because they are less cautious due to less fear, and so this is a secondary measure.
Time before needing a break or quitting the virtual reality plank walk | 1 hour after taking acetaminophen or placebo
  (Unless there are ceiling effects in which >90% of participants do not quit early or need a break). Amount of time before a participant takes their headset off early, to quit or for a break, due to being overwhelmed.

CONTACTS AND LOCATIONS:
Overall Officials: Pat Barclay, Ph.D., Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Open Science Framework
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon publication or within two years
Access Criteria: Open Access
URL: https://osf.io/ma3ur/?view_only=a9ed5d5d09f24277a66efbf46f24d31f